CLINICAL TRIAL: NCT04384107
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active-Comparator-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 in Healthy Japanese Infants
Brief Title: Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 in Healthy Japanese Infants (V114-033)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-033; V114-033 (Other: Merck); 205287 (Registry Identifier: JAPIC-CTI); 2019-003644-68 (EudraCT Number)
Record Dates: First submitted 2020-05-11; First posted 2020-05-12 (Actual); Results first posted 2022-11-15 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- V114 (Experimental): Participants will receive a single 0.5 mL subcutaneous injection of V114 administered at 2 to 6 months of age, and second and third dose is administered at an interval of ≥27 days from the prior dose. The fourth dose is administered at 12 to 15 months of age.
  Interventions: Biological: V114
- Pneumococcal 13-valent Conjugate Vaccine (PCV13) (Active Comparator): Participants will receive a single 0.5 mL subcutaneous injection of PCV13 administered at 2 to 6 months of age, and second and third dose is administered at an interval of ≥27 days from the prior dose. The fourth dose is administered at 12 to 15 months of age.
  Interventions: Biological: PCV13

INTERVENTIONS:
Biological: V114 — 15-valent pneumococcal conjugate vaccine containing 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) present in PCV13 plus 2 additional serotypes (22F, 33F) in each subcutaneous 0.5 mL single dose.
  Other Names: VAXNEUVANCE™; Pneumococcal 15-Valent Conjugate Vaccine
  Arms: V114
Biological: PCV13 — 13-valent pneumococcal conjugate vaccine containing 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) in each subcutaneous 0.5 mL single dose.
  Other Names: Prevnar 13™
  Arms: Pneumococcal 13-valent Conjugate Vaccine (PCV13)

SUMMARY:
The purpose of this clinical study is to evaluate the safety and immunogenicity of a 4-dose schedule (3-dose primary series followed by a toddler dose) of V114 compared with Pneumococcal 13-valent Conjugate Vaccine (PCV13). The hypotheses are that: 1) V114 is non-inferior to PCV13 for the 13 shared serotypes between V114 and PCV13 based on the response rates at 30 days following dose 3; 2) V114 is non-inferior to PCV13 for the 2 unique V114 serotypes based on the response rate of the 2 unique V114 serotypes at 30 days following dose 3; 3) V114 is non-inferior to PCV13 for the 13 shared serotypes between V114 and PCV13 based on anti-pneumococcal polysaccharide (PnPs) serotype-specific Immunoglobulin G (IgG) geometric mean concentrations (GMCs) at 30 days following dose 3.

ELIGIBILITY:
Inclusion Criteria:

- Japanese male or female

Exclusion Criteria:

* Has a history of invasive pneumococcal disease (IPD)
* Has a known hypersensitivity to any component of the pneumococcal conjugate vaccine (PCV), or any diphtheria toxoid containing vaccine
* Has a known or suspected impairment of immunological function
* Has a history of congenital or acquired immunodeficiency
* Has or his/her mother has a documented human immunodeficiency virus (HIV) infection
* Has or his/her mother has a documented hepatitis B surface antigen-positive test
* Has known or history of functional or anatomic asplenia
* Has a history of autoimmune disease
* Has a known neurologic or cognitive behavioral disorder
* Has received a dose of any pneumococcal vaccine prior to study entry
* Has received a blood transfusion or blood products, including immunoglobulins

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 694 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (45):
- Japan (45):
  - Morinaga Maternity Clinic ( Site 3345), Kasugai, Aichi-ken
  - Social Medical Corporation Koujunkai Daido Clinic ( Site 3326), Nagoya, Aichi-ken
  - Kyoritsu Narashinodai Hospital ( Site 3332), Funabashi, Chiba
  - Sotobo Children's Clinic ( Site 3323), Isumi, Chiba
  - Yokoyama Children's Clinic ( Site 3309), Kasuga, Fukuoka
  - Chugoku Rosai Hospital ( Site 3340), Kure, Hiroshima
  - Tsuchiura Kyodo General Hospital ( Site 3327), Tsuchiura, Ibaraki
  - Kagoshima Children's Hospital ( Site 3342), Hioki, Kagoshima-ken
  - Kawasaki Municipal Hospital ( Site 3302), Kawasaki, Kanagawa
  - National Hospital Organization Sagamihara National Hospital ( Site 3303), Sagamihara, Kanagawa
  - JOHAS Yokohama Rosai Hospital ( Site 3343), Yokohama, Kanagawa
  - National Hospital Organization Mie Chuo Medical Center ( Site 3308), Tsu, Mie-ken
  - National Hospital Organization Sendai Medical Center ( Site 3311), Sendai, Miyagi
  - Ina Central Hospital ( Site 3346), Ina, Nagano
  - Aizawa Hospital ( Site 3313), Matsumoto, Nagano
  - Taniguchi Hospital ( Site 3310), Izumisano, Osaka
  - Medical corporation Waffle GunGunkids Clinic ( Site 3329), Sakai, Osaka
  - Suita Municipal Hospital ( Site 3338), Suita, Osaka
  - Takatsuki General Hospital ( Site 3318), Takatsuki, Osaka
  - Aiwa Hospital ( Site 3336), Kawagoe, Saitama
  - Saiseikai Kawaguchi General Hospital ( Site 3304), Kawaguchi, Saitama
  - Hara Children's Clinic ( Site 3339), Tokorozawa, Saitama
  - National Hospital Organization Saitama Hospital ( Site 3312), Wako, Saitama
  - Saiseikai Shiga Hospital ( Site 3349), Rittō, Shiga
  - Kobayashi Pediatric Clinic ( Site 3301), Fujieda, Shizuoka
  - Saiwai Kodomo Clinic ( Site 3331), Tachikawa, Tokyo
  - Nishida Kodomo Clinic ( Site 3306), Tama, Tokyo
  - Fukui Aiiku Hospital ( Site 3315), Fukui
  - Fukui-ken Saiseikai Hospital ( Site 3314), Fukui
  - Shindo Children's Clinic ( Site 3325), Fukuoka
  - Kurokawa Michiko Pediatric Clinic ( Site 3319), Fukuoka
  - Shimomura Pediatrics Clinic ( Site 3320), Fukuoka
  - INAMITSU Children's Clinic ( Site 3321), Fukuoka
  - Nagamine Soyokaze Clinic ( Site 3348), Kumamoto
  - Minaminagano Medical Center Shinonoi General Hospital ( Site 3344), Nagano
  - Saiseikai Noe Hospital ( Site 3330), Osaka
  - Kubota Children's Clinic ( Site 3334), Osaka
  - Sano Kids Clinic ( Site 3341), Osaka
  - Aizenbashi Hospital ( Site 3317), Osaka
  - Japanese Red Cross Shizuoka Hospital ( Site 3322), Shizuoka
  - Shizuoka City Shimizu Hospital ( Site 3347), Shizuoka
  - Hosaka Children's Clinic ( Site 3307), Tokyo
  - The Fraternity Memorial Hospital ( Site 3333), Tokyo
  - Okawa Children & Family Clinic ( Site 3305), Tokyo
  - Toyama City Hospital ( Site 3328), Toyama

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Suzuki H, Fujita H, Iwai K, Kuroki H, Taniyama K, Shizuya T, Kishino H, Igarashi R, Shirakawa M, Sawata M. Safety and immunogenicity of 15-valent pneumococcal conjugate vaccine in Japanese healthy infants: A phase III study (V114-033). Vaccine. 2023 Jul 31;41(34):4933-4940. doi: 10.1016/j.vaccine.2023.05.064. Epub 2023 Jun 19. PMID 37344262

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled healthy Japanese infants at 2 to 6 months of age.
Pre-assignment Details: 694 infants were randomized in a 1:1 ratio with stratification into 3 categories by age category (2 months, 3 months and 4 to 6 months of age), to receive either V114 or Pneumococcal 13-valent Conjugate Vaccine (PCV13).
Groups:
- V114: Participants received a single 0.5 ml subcutaneous injection of V114 administered at 2 to 6 months of age, and second and third dose is administered at an interval of ≥27 days from the prior dose. The fourth dose is administered at 12 to 15 months of age.
- PCV13: Participants received a single 0.5 mL subcutaneous injection of PCV13 administered at 2 to 6 months of age, and second and third dose is administered at an interval of ≥27 days from the prior dose. The fourth dose is administered at 12 to 15 months of age.
Period: Overall Study
Arm/Group | V114 | PCV13
Started | 347 | 347
Dose 1 | 347 | 346
Dose 2 | 344 | 346
Dose 3 | 343 | 346
Dose 4 | 340 | 342
Completed | 338 | 341
Not Completed | 9 | 6
Not completed — Withdrawal By Parent/Guardian | 8 | 6
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 | PCV13 | Total
Number analyzed (Participants) | 347 | 347 | 694
Age, Continuous [Mean (Standard Deviation); unit: months] | 2.4 (0.4) | 2.4 (0.4) | 2.4 (0.4)
Age, Customized [Count of Participants; unit: Participants]
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 347 | 347 | 694
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 173 | 339
  Male | 181 | 174 | 355
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 347 | 347 | 694
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 347 | 347 | 694
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-Site Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following any injection with either V114 or PCV13 the percentage of participants with solicited injection-site AEs was assessed. The solicited injection-site AEs were erythema, induration, pain, and swelling.
Time Frame: Day 1 to Day 14 post any vaccination, up to a total of 13.5 months
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | PCV13
Number analyzed (Participants) | 347 | 346
Percentage of Participants
  Injection site erythema | 88.2 | 89.3
  Injection site induration | 81.0 | 81.2
  Injection site pain | 31.1 | 24.0
  Injection site swelling | 75.8 | 79.8
Statistical Analysis 1: Comparison: V114 vs PCV13; Injection site erythema; Test type: Other — Estimated differences, confidence intervals (CIs), and p-values are calculated based on the Miettinen & Nurminen method and are provided in accordance with the statistical analysis plan; p = 0.641, Miettinen & Nurminen; Difference in Percent = -1.1, 95% CI 2-sided [-5.9 to 3.6]
Statistical Analysis 2: Comparison: V114 vs PCV13; Injection site induration; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.937, Miettinen & Nurminen; Difference in Percent = -0.2, 95% CI 2-sided [-6.1 to 5.6]
Statistical Analysis 3: Comparison: V114 vs PCV13; Injection site pain; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.036, Miettinen & Nurminen; Difference in Percent = 7.1, 95% CI 2-sided [0.5 to 13.8]
Statistical Analysis 4: Comparison: V114 vs PCV13; Injection site swelling; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.208, Miettinen & Nurminen; Difference in Percent = -4.0, 95% CI 2-sided [-10.2 to 2.2]

2. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Following any of the injections with either V114 or PCV13, the percentage of participants with solicited systemic AEs was assessed. The solicited systemic AEs assessed were decreased appetite, irritability, somnolence, and urticaria.
Time Frame: Day 1 to Day 14 post any vaccination, up to a total of 13.5 months
Population: All randomized participants who received at least 1 dose of study vaccination were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | PCV13
Number analyzed (Participants) | 347 | 346
Percentage of Participants
  Decreased appetite | 23.9 | 24.3
  Irritability | 66.6 | 60.7
  Somnolence | 55.9 | 54.9
  Urticaria | 4.0 | 4.3
Statistical Analysis 1: Comparison: V114 vs PCV13; Decreased appetite; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.912, Miettinen & Nurminen; Difference in Percent = -0.4, 95% CI 2-sided [-6.7 to 6.0]
Statistical Analysis 2: Comparison: V114 vs PCV13; Irritability; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.108, Miettinen & Nurminen; Difference in Percent = 5.9, 95% CI 2-sided [-1.3 to 13.0]
Statistical Analysis 3: Comparison: V114 vs PCV13; Somnolence; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.792, Miettinen & Nurminen; Difference in Percent = 1.0, 95% CI 2-sided [-6.4 to 8.4]
Statistical Analysis 4: Comparison: V114 vs PCV13; Urticaria; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.843, Miettinen & Nurminen; Difference in Percent = -0.3, 95% CI 2-sided [-3.5 to 2.8]

3. Primary Outcome: Percentage of Participants With Vaccine-Related Serious Adverse Events
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. The percentage of participants with a vaccine-related SAE following dose 1 (with either V114 or PCV13) was reported. Vaccine-related SAEs were counted starting after vaccine dose 1 through completion of study.
Time Frame: ~1 month after Dose 4, up to a total of 14 months
Population: All randomized participants who received at least 1 dose of the relevant study vaccination for the timepoint of interest were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | PCV13
Number analyzed (Participants) | 347 | 346
Percentage of Participants | 0.3 | 0.3
Statistical Analysis 1: Comparison: V114 vs PCV13; Test type: Other — Estimated differences and CIs are calculated based on the Miettinen & Nurminen method and are provided in accordance with the statistical analysis plan; Difference in Percent = -0.0, 95% CI 2-sided [-1.4 to 1.3]

4. Primary Outcome: Percentage of Participants Meeting the Serotype Specific Immunoglobulin G Threshold Value of ≥0.35 μg/mL for Each Serotype in V114 After Dose 3
Description: The anti-pneumococcal polysaccharide (PnPs) serotype-specific immunoglobulin G (IgG) response rates (percentage of participants meeting serotype-specific IgG threshold value of ≥0.35 μg/mL of participants administered V114 versus participants administered PCV13) for the 15 serotypes contained in V114 were determined using an electrochemiluminescence assay.
Time Frame: 30 Days after Dose 3, up to a total of 11 months
Population: All randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity outcome measure and who had sufficient data to perform the analyses were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | PCV13
Number analyzed (Participants) | 339 | 343
Percentage of Participants
  Serotype 1 (Shared) | 99.7 | 100.0
  Serotype 3 (Shared) | 100.0 | 97.7
  Serotype 4 (Shared) | 100.0 | 100.0
  Serotype 5 (Shared): number analyzed (Participants) | 338 | 343
  Serotype 5 (Shared) | 98.8 | 100.0
  Serotype 6A (Shared) | 99.1 | 100.0
  Serotype 6B (Shared) | 95.0 | 98.8
  Serotype 7F (Shared) | 99.7 | 100.0
  Serotype 9V (Shared) | 99.7 | 100.0
  Serotype 14 (Shared): number analyzed (Participants) | 339 | 342
  Serotype 14 (Shared) | 99.4 | 99.7
  Serotype 18C (Shared) | 98.8 | 100.0
  Serotype 19A (Shared) | 99.7 | 100.0
  Serotype 19F (Shared) | 100.0 | 100.0
  Serotype 23F (Shared): number analyzed (Participants) | 338 | 342
  Serotype 23F (Shared) | 97.9 | 99.7
  Serotype 22F (Unique to V114) | 99.7 | NA — This analysis represents the difference between response rate to Serotype 22F in recipients of V114 and lowest response (Serotype 3 at 97.7) in recipients of PCV13 for shared serotypes.
  Serotype 33F (Unique to V114) | 90.9 | NA — This analysis represents the difference between response rate to Serotype 33F in recipients of V114 and lowest response (Serotype 3 at 97.7) in recipients of PCV13 for shared serotypes.
Statistical Analysis 1: Comparison: V114 vs PCV13; Serotype 1: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — The stratum-adjusted proportion difference using the Cochran-Mantel-Haenszel weight, and the corresponding 95% CI and p-value based on the method of Miettinen and Nurminen stratified by age category. A conclusion of non-inferiority of V114 to PCV13 is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - PCV13) being >-10 percentage points (1-sided p-value <0.025); p < 0.001, Miettinen and Nurminen; Difference in Percent = -0.3, 95% CI 2-sided [-1.7 to 0.8]
Statistical Analysis 2: Comparison: V114 vs PCV13; Serotype 3: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = 2.3, 95% CI 2-sided [1.0 to 4.5]
Statistical Analysis 3: Comparison: V114 vs PCV13; Serotype 4: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 4: Comparison: V114 vs PCV13; Serotype 5: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = -1.2, 95% CI 2-sided [-3.0 to -0.1]
Statistical Analysis 5: Comparison: V114 vs PCV13; Serotype 6A: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = -0.9, 95% CI 2-sided [-2.6 to 0.2]
Statistical Analysis 6: Comparison: V114 vs PCV13; Serotype 6B: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = -3.9, 95% CI 2-sided [-6.9 to -1.3]
Statistical Analysis 7: Comparison: V114 vs PCV13; Serotype 7F: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = -0.3, 95% CI 2-sided [-1.7 to 0.8]
Statistical Analysis 8: Comparison: V114 vs PCV13; Serotype 9V: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = -0.3, 95% CI 2-sided [-1.7 to 0.8]
Statistical Analysis 9: Comparison: V114 vs PCV13; Serotype 14: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = -0.3, 95% CI 2-sided [-1.9 to 1.1]
Statistical Analysis 10: Comparison: V114 vs PCV13; Serotype 18C: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = -1.2, 95% CI 2-sided [-3.0 to -0.1]
Statistical Analysis 11: Comparison: V114 vs PCV13; Serotype 19A: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = -0.3, 95% CI 2-sided [-1.7 to 0.8]
Statistical Analysis 12: Comparison: V114 vs PCV13; Serotype 19F: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 13: Comparison: V114 vs PCV13; Serotype 23F: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = -1.8, 95% CI 2-sided [-4.0 to -0.2]
Statistical Analysis 14: Comparison: V114 vs PCV13; Serotype 22F: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percent = 2.0, 95% CI 2-sided [0.4 to 4.3]
Statistical Analysis 15: Comparison: V114 vs PCV13; Serotype 33F: Participants With IgG ≥0.35 μg/mL; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.048, Miettinen and Nurminen; Difference in Percent = -6.8, 95% CI 2-sided [-10.6 to -3.5]

5. Primary Outcome: Geometric Mean Concentration of Serotype-Specific IgG for the 13 Shared Serotypes in V114 and PCV13 After Dose 3
Description: The anti-PnPs serotype-specific IgG Geometric Mean Concentrations (GMCs) of participants administered V114 versus participants administered PCV13 for the 13 serotypes shared in V114 and PCV13 were determined using an electrochemiluminescence assay.
Time Frame: 30 Days after Dose 3, up to a total of 11 months
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | PCV13
Number analyzed (Participants) | 339 | 343
μg/mL
  Serotype 1 (Shared) | 2.39 [2.19 to 2.62] | 3.95 [3.61 to 4.32]
  Serotype 3 (Shared) | 2.63 [2.39 to 2.89] | 1.42 [1.29 to 1.56]
  Serotype 4 (Shared) | 2.98 [2.71 to 3.27] | 3.54 [3.23 to 3.89]
  Serotype 5 (Shared): number analyzed (Participants) | 338 | 343
  Serotype 5 (Shared) | 2.59 [2.32 to 2.89] | 3.35 [3.00 to 3.74]
  Serotype 6A (Shared) | 2.51 [2.26 to 2.79] | 4.45 [4.00 to 4.94]
  Serotype 6B (Shared) | 2.46 [2.14 to 2.82] | 4.17 [3.63 to 4.79]
  Serotype 7F (Shared) | 4.38 [3.95 to 4.85] | 5.22 [4.71 to 5.78]
  Serotype 9V (Shared) | 3.09 [2.80 to 3.41] | 3.55 [3.22 to 3.92]
  Serotype 14 (Shared): number analyzed (Participants) | 339 | 342
  Serotype 14 (Shared) | 8.99 [7.96 to 10.14] | 12.03 [10.66 to 13.57]
  Serotype 18C (Shared) | 2.85 [2.58 to 3.14] | 3.85 [3.49 to 4.25]
  Serotype 19A (Shared) | 3.44 [3.14 to 3.77] | 5.28 [4.82 to 5.79]
  Serotype 19F (Shared) | 4.24 [3.93 to 4.58] | 5.65 [5.24 to 6.10]
  Serotype 23F (Shared): number analyzed (Participants) | 338 | 342
  Serotype 23F (Shared) | 2.42 [2.15 to 2.72] | 2.95 [2.62 to 3.32]
Statistical Analysis 1: Comparison: V114 vs PCV13; Serotype 1: IgG GMC Ratio; Test type: Non-Inferiority — Based on a linear model with natural log-transformed IgG concentrations as response variable, and vaccination group and age category as factors. A conclusion of non-inferiority of V114 to PCV13 is based on the lower bound of the 2-sided 95% CI for the GMC ratio (V114/PCV13) being >0.5 (1-sided p-value <0.025); p < 0.001, Linear model; GMC Ratio = 0.61, 95% CI 2-sided [0.55 to 0.67]
Statistical Analysis 2: Comparison: V114 vs PCV13; Serotype 3: IgG GMC Ratio; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Linear model; GMC Ratio = 1.85, 95% CI 2-sided [1.67 to 2.05]
Statistical Analysis 3: Comparison: V114 vs PCV13; Serotype 4: IgG GMC Ratio; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Linear model; GMC Ratio = 0.84, 95% CI 2-sided [0.76 to 0.93]
Statistical Analysis 4: Comparison: V114 vs PCV13; Serotype 5: IgG GMC Ratio; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Linear model; GMC Ratio = 0.77, 95% CI 2-sided [0.69 to 0.87]
Statistical Analysis 5: Comparison: V114 vs PCV13; Serotype 6A: IgG GMC Ratio; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p = 0.019, Linear model; GMC Ratio = 0.56, 95% CI 2-sided [0.50 to 0.63]
Statistical Analysis 6: Comparison: V114 vs PCV13; Serotype 6B: IgG GMC Ratio; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p = 0.015, Linear model; GMC Ratio = 0.59, 95% CI 2-sided [0.51 to 0.68]
Statistical Analysis 7: Comparison: V114 vs PCV13; Serotype 7F: IgG GMC Ratio; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Linear model; GMC Ratio = 0.84, 95% CI 2-sided [0.75 to 0.94]
Statistical Analysis 8: Comparison: V114 vs PCV13; Serotype 9V: IgG GMC Ratio; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Linear model; GMC Ratio = 0.87, 95% CI 2-sided [0.78 to 0.97]
Statistical Analysis 9: Comparison: V114 vs PCV13; Serotype 14: IgG GMC Ratio; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Linear model; GMC Ratio = 0.75, 95% CI 2-sided [0.66 to 0.85]
Statistical Analysis 10: Comparison: V114 vs PCV13; Serotype 18C: IgG GMC Ratio; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Linear model; GMC Ratio = 0.74, 95% CI 2-sided [0.67 to 0.82]
Statistical Analysis 11: Comparison: V114 vs PCV13; Serotype 19A: IgG GMC Ratio; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Linear model; GMC Ratio = 0.65, 95% CI 2-sided [0.59 to 0.72]
Statistical Analysis 12: Comparison: V114 vs PCV13; Serotype 19F: IgG GMC Ratio; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Linear model; GMC Ratio = 0.75, 95% CI 2-sided [0.69 to 0.82]

6. Secondary Outcome: GMC of Serotype-Specific IgG for the 2 Unique V114 Serotypes After Dose 3
Description: The anti-PnPs serotype-specific IgG GMCs of participants administered V114 versus participants administered PCV13 for the 2 unique V114 serotypes was determined using an electrochemiluminescence assay.
Time Frame: 30 days after Dose 3, up to a total of 11 months
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | PCV13
Number analyzed (Participants) | 339 | 343
μg/mL
  Serotype 22F (Unique to V114) | 6.59 [5.95 to 7.30] | 0.06 [0.06 to 0.07]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 339 | 337
  Serotype 33F (Unique to V114) | 1.85 [1.60 to 2.14] | 0.06 [0.05 to 0.07]
Statistical Analysis 1: Comparison: V114 vs PCV13; Serotype 22F: IgG GMC Ratio; Test type: Other — Based on a linear model with natural log-transformed IgG concentrations as response variable, and vaccination group and age category as factors; GMC Ratio = 107.45, 95% CI 2-sided [96.18 to 120.03]
Statistical Analysis 2: Comparison: V114 vs PCV13; Serotype 33F: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 32.48, 95% CI 2-sided [27.72 to 38.05]

7. Secondary Outcome: Percentage of Participants Meeting the Serotype Specific IgG Threshold Value of ≥0.35 μg/mL for Each Serotype in V114 After Dose 4
Description: The anti-PnPs serotype-specific IgG response rates (percentage of participants meeting serotype-specific IgG threshold value of ≥0.35 μg/mL of participants administered V114 versus participants administered PCV13) for the 15 serotypes contained in V114 were determined using an electrochemiluminescence assay.
Time Frame: 30 Days after Dose 4, up to a total of 14 months
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 | PCV13
Number analyzed (Participants) | 333 | 334
Percentage of Participants
  Serotype 1 (Shared) | 99.7 | 100.0
  Serotype 3 (Shared) | 100.0 | 96.7
  Serotype 4 (Shared) | 99.7 | 100.0
  Serotype 5 (Shared) | 100.0 | 100.0
  Serotype 6A (Shared) | 100.0 | 100.0
  Serotype 6B (Shared) | 100.0 | 100.0
  Serotype 7F (Shared) | 100.0 | 100.0
  Serotype 9V (Shared) | 100.0 | 100.0
  Serotype 14 (Shared) | 100.0 | 100.0
  Serotype 18C (Shared) | 100.0 | 100.0
  Serotype 19A (Shared) | 100.0 | 100.0
  Serotype 19F (Shared) | 100.0 | 100.0
  Serotype 23F (Shared): number analyzed (Participants) | 332 | 334
  Serotype 23F (Shared) | 99.7 | 99.4
  Serotype 22F (Unique to V114): number analyzed (Participants) | 333 | 327
  Serotype 22F (Unique to V114) | 100.0 | 5.2
  Serotype 33F (Unique to V114): number analyzed (Participants) | 333 | 313
  Serotype 33F (Unique to V114) | 100.0 | 11.5
Statistical Analysis 1: Comparison: V114 vs PCV13; Serotype 1: Participants With IgG ≥0.35 μg/mL; Test type: Other — The stratum-adjusted proportion difference using the Cochran-Mantel-Haenszel weight, and the corresponding 95% CI based on the method of Miettinen and Nurminen stratified by age category; Difference in Percent = -0.3, 95% CI 2-sided [-1.7 to 0.8]
Statistical Analysis 2: Comparison: V114 vs PCV13; Serotype 3: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 3.3, 95% CI 2-sided [1.8 to 5.8]
Statistical Analysis 3: Comparison: V114 vs PCV13; Serotype 4: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = -0.3, 95% CI 2-sided [-1.7 to 0.8]
Statistical Analysis 4: Comparison: V114 vs PCV13; Serotype 5: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 5: Comparison: V114 vs PCV13; Serotype 6A: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 6: Comparison: V114 vs PCV13; Serotype 6B: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 7: Comparison: V114 vs PCV13; Serotype 7F: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 8: Comparison: V114 vs PCV13; Serotype 9V: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 9: Comparison: V114 vs PCV13; Serotype 14: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 10: Comparison: V114 vs PCV13; Serotype 18C: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 11: Comparison: V114 vs PCV13; Serotype 19A: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 12: Comparison: V114 vs PCV13; Serotype 19F: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 0.0, 95% CI 2-sided [-1.1 to 1.1]
Statistical Analysis 13: Comparison: V114 vs PCV13; Serotype 23F: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 0.3, 95% CI 2-sided [-1.1 to 1.9]
Statistical Analysis 14: Comparison: V114 vs PCV13; Serotype 22F: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 94.8, 95% CI 2-sided [91.8 to 96.7]
Statistical Analysis 15: Comparison: V114 vs PCV13; Serotype 33F: Participants With IgG ≥0.35 μg/mL; Test type: Other — [test comment as in outcome 7, analysis 1]; Difference in Percent = 88.5, 95% CI 2-sided [84.5 to 91.6]

8. Secondary Outcome: GMC of Serotype-Specific IgG for Each Serotype in V114 After Dose 4
Description: The anti-PnPs serotype-specific IgG GMCs of participants administered V114 versus participants administered PCV13 for the 15 serotypes contained in V114 was determined using an electrochemiluminescence assay.
Time Frame: 30 Days after Dose 4, up to a total of 14 months
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | PCV13
Number analyzed (Participants) | 333 | 334
μg/mL
  Serotype 1 (Shared) | 2.74 [2.47 to 3.04] | 5.19 [4.68 to 5.77]
  Serotype 3 (Shared) | 2.18 [1.97 to 2.41] | 1.28 [1.15 to 1.41]
  Serotype 4 (Shared) | 2.91 [2.57 to 3.30] | 3.18 [2.81 to 3.59]
  Serotype 5 (Shared) | 4.43 [3.96 to 4.95] | 6.65 [5.95 to 7.43]
  Serotype 6A (Shared) | 6.05 [5.36 to 6.81] | 9.41 [8.35 to 10.60]
  Serotype 6B (Shared) | 8.03 [7.12 to 9.05] | 10.88 [9.66 to 12.26]
  Serotype 7F (Shared) | 5.80 [5.15 to 6.54] | 7.15 [6.35 to 8.05]
  Serotype 9V (Shared) | 4.27 [3.79 to 4.81] | 5.18 [4.60 to 5.83]
  Serotype 14 (Shared) | 9.51 [8.45 to 10.69] | 11.26 [10.02 to 12.66]
  Serotype 18C (Shared) | 5.21 [4.60 to 5.89] | 5.21 [4.61 to 5.90]
  Serotype 19A (Shared) | 6.88 [6.20 to 7.63] | 8.37 [7.55 to 9.28]
  Serotype 19F (Shared) | 6.53 [5.89 to 7.22] | 7.76 [7.01 to 8.58]
  Serotype 23F (Shared): number analyzed (Participants) | 332 | 334
  Serotype 23F (Shared) | 3.75 [3.26 to 4.31] | 6.22 [5.42 to 7.15]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 333 | 327
  Serotype 22F (Unique to V114) | 11.42 [10.31 to 12.66] | 0.13 [0.12 to 0.15]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 333 | 313
  Serotype 33F (Unique to V114) | 6.14 [5.48 to 6.89] | 0.14 [0.12 to 0.15]
Statistical Analysis 1: Comparison: V114 vs PCV13; Serotype 1: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 0.53, 95% CI 2-sided [0.47 to 0.59]
Statistical Analysis 2: Comparison: V114 vs PCV13; Serotype 3: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 1.71, 95% CI 2-sided [1.53 to 1.90]
Statistical Analysis 3: Comparison: V114 vs PCV13; Serotype 4: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 0.92, 95% CI 2-sided [0.80 to 1.05]
Statistical Analysis 4: Comparison: V114 vs PCV13; Serotype 5: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 0.67, 95% CI 2-sided [0.59 to 0.75]
Statistical Analysis 5: Comparison: V114 vs PCV13; Serotype 6A: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 0.64, 95% CI 2-sided [0.56 to 0.73]
Statistical Analysis 6: Comparison: V114 vs PCV13; Serotype 6B: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 0.74, 95% CI 2-sided [0.65 to 0.84]
Statistical Analysis 7: Comparison: V114 vs PCV13; Serotype 7F: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 0.81, 95% CI 2-sided [0.71 to 0.92]
Statistical Analysis 8: Comparison: V114 vs PCV13; Serotype 9V: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 0.83, 95% CI 2-sided [0.73 to 0.94]
Statistical Analysis 9: Comparison: V114 vs PCV13; Serotype 14: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 0.84, 95% CI 2-sided [0.74 to 0.96]
Statistical Analysis 10: Comparison: V114 vs PCV13; Serotype 18C: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 1.00, 95% CI 2-sided [0.87 to 1.14]
Statistical Analysis 11: Comparison: V114 vs PCV13; Serotype 19A: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 0.82, 95% CI 2-sided [0.73 to 0.92]
Statistical Analysis 12: Comparison: V114 vs PCV13; Serotype 19F: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 0.84, 95% CI 2-sided [0.75 to 0.94]
Statistical Analysis 13: Comparison: V114 vs PCV13; Serotype 23F: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 0.60, 95% CI 2-sided [0.52 to 0.70]
Statistical Analysis 14: Comparison: V114 vs PCV13; Serotype 22F: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 86.74, 95% CI 2-sided [77.61 to 96.95]
Statistical Analysis 15: Comparison: V114 vs PCV13; Serotype 33F: IgG GMC Ratio; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC Ratio = 45.44, 95% CI 2-sided [40.07 to 51.54]

9. Secondary Outcome: Geometric Mean Titer of Serotype-Specific Opsonophagocytic Activity for Each Serotype in V114 After Dose 3
Description: The anti-PnPs serotype-specific opsonophagocytic activity (OPA) and geometric mean titers (GMTs) of participants administered V114 versus participants administered PCV13 for the 15 serotypes contained in V114 was determined using a multiplexed opsonophagocytic assay.
Time Frame: 30 Days after Dose 3, up to a total of 11 months
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V114 | PCV13
Number analyzed (Participants) | 337 | 340
Titer
  Serotype 1 (Shared): number analyzed (Participants) | 336 | 340
  Serotype 1 (Shared) | 211.51 [180.48 to 247.86] | 322.44 [275.23 to 377.76]
  Serotype 3 (Shared): number analyzed (Participants) | 333 | 336
  Serotype 3 (Shared) | 660.68 [586.60 to 744.11] | 471.43 [418.48 to 531.08]
  Serotype 4 (Shared): number analyzed (Participants) | 334 | 338
  Serotype 4 (Shared) | 3984.87 [3537.66 to 4488.62] | 4118.16 [3656.82 to 4637.70]
  Serotype 5 (Shared): number analyzed (Participants) | 336 | 339
  Serotype 5 (Shared) | 1241.69 [1098.82 to 1403.14] | 1358.43 [1202.35 to 1534.79]
  Serotype 6A (Shared): number analyzed (Participants) | 334 | 336
  Serotype 6A (Shared) | 9124.96 [7894.53 to 10547.16] | 11956.64 [10340.85 to 13824.91]
  Serotype 6B (Shared): number analyzed (Participants) | 334 | 338
  Serotype 6B (Shared) | 8416.19 [7243.92 to 9778.18] | 10421.94 [8972.87 to 12105.02]
  Serotype 7F (Shared): number analyzed (Participants) | 334 | 338
  Serotype 7F (Shared) | 22324.41 [19365.68 to 25735.19] | 27396.28 [23771.84 to 31573.33]
  Serotype 9V (Shared): number analyzed (Participants) | 334 | 338
  Serotype 9V (Shared) | 2725.29 [2399.27 to 3095.62] | 3338.40 [2939.75 to 3791.11]
  Serotype 14 (Shared): number analyzed (Participants) | 334 | 339
  Serotype 14 (Shared) | 14175.13 [12024.73 to 16710.08] | 12288.35 [10433.90 to 14472.40]
  Serotype 18C (Shared): number analyzed (Participants) | 334 | 339
  Serotype 18C (Shared) | 3698.24 [3346.73 to 4086.66] | 3705.21 [3353.84 to 4093.39]
  Serotype 19A (Shared): number analyzed (Participants) | 335 | 339
  Serotype 19A (Shared) | 2709.90 [2418.02 to 3037.02] | 3961.10 [3535.23 to 4438.26]
  Serotype 19F (Shared): number analyzed (Participants) | 334 | 339
  Serotype 19F (Shared) | 2371.39 [2141.38 to 2624.87] | 2541.27 [2297.18 to 2811.29]
  Serotype 23F (Shared): number analyzed (Participants) | 334 | 340
  Serotype 23F (Shared) | 11861.63 [10118.30 to 13905.32] | 18957.26 [16186.86 to 22201.82]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 333 | 333
  Serotype 22F (Unique to V114) | 5575.08 [4769.68 to 6516.47] | 9.95 [8.51 to 11.63]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 333 | 334
  Serotype 33F (Unique to V114) | 23888.79 [17632.59 to 32364.75] | 121.79 [89.73 to 165.32]
Statistical Analysis 1: Comparison: V114 vs PCV13; Serotype 1: OPA GMT Ratio; Test type: Other — Based on a linear model with natural log-transformed OPA titers as response variable, and vaccination group and age category as factors; GMT Ratio = 0.66, 95% CI 2-sided [0.55 to 0.78]
Statistical Analysis 2: Comparison: V114 vs PCV13; Serotype 3: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 1.40, 95% CI 2-sided [1.23 to 1.59]
Statistical Analysis 3: Comparison: V114 vs PCV13; Serotype 4: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.97, 95% CI 2-sided [0.85 to 1.10]
Statistical Analysis 4: Comparison: V114 vs PCV13; Serotype 5: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.91, 95% CI 2-sided [0.80 to 1.04]
Statistical Analysis 5: Comparison: V114 vs PCV13; Serotype 6A: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.76, 95% CI 2-sided [0.65 to 0.89]
Statistical Analysis 6: Comparison: V114 vs PCV13; Serotype 6B: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 0.81, 95% CI 2-sided [0.69 to 0.95]
Statistical Analysis 7: Comparison: V114 vs PCV13; Serotype 7F: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMC Ratio = 0.81, 95% CI 2-sided [0.70 to 0.95]
Statistical Analysis 8: Comparison: V114 vs PCV13; Serotype 9V: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.82, 95% CI 2-sided [0.71 to 0.94]
Statistical Analysis 9: Comparison: V114 vs PCV13; Serotype 14: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 1.15, 95% CI 2-sided [0.97 to 1.38]
Statistical Analysis 10: Comparison: V114 vs PCV13; Serotype 18C: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 1.00, 95% CI 2-sided [0.90 to 1.11]
Statistical Analysis 11: Comparison: V114 vs PCV13; Serotype 19A: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.68, 95% CI 2-sided [0.61 to 0.77]
Statistical Analysis 12: Comparison: V114 vs PCV13; Serotype 19F: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.93, 95% CI 2-sided [0.84 to 1.04]
Statistical Analysis 13: Comparison: V114 vs PCV13; Serotype 23F: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.63, 95% CI 2-sided [0.53 to 0.74]
Statistical Analysis 14: Comparison: V114 vs PCV13; Serotype 22F: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 560.46, 95% CI 2-sided [474.05 to 662.63]
Statistical Analysis 15: Comparison: V114 vs PCV13; Serotype 33F: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 196.14, 95% CI 2-sided [141.85 to 271.21]

10. Secondary Outcome: GMT of Serotype-Specific OPA for Each Serotype in V114 After Dose 4
Description: as for outcome 9
Time Frame: 30 Days after Dose 4, up to a total of 14 months
Population: The first 50% of all participants with sufficient serum volume after dose 3 to evaluate OPA responses were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V114 | PCV13
Number analyzed (Participants) | 157 | 156
Titer
  Serotype 1 (Shared): number analyzed (Participants) | 156 | 156
  Serotype 1 (Shared) | 453.42 [327.21 to 628.32] | 854.50 [616.64 to 1184.10]
  Serotype 3 (Shared): number analyzed (Participants) | 150 | 146
  Serotype 3 (Shared) | 1444.00 [1166.36 to 1787.72] | 893.97 [720.25 to 1109.58]
  Serotype 4 (Shared): number analyzed (Participants) | 153 | 152
  Serotype 4 (Shared) | 4531.52 [3592.99 to 5715.21] | 6264.94 [4957.63 to 7916.97]
  Serotype 5 (Shared): number analyzed (Participants) | 157 | 154
  Serotype 5 (Shared) | 1853.08 [1439.01 to 2386.30] | 2151.95 [1669.81 to 2773.30]
  Serotype 6A (Shared): number analyzed (Participants) | 152 | 152
  Serotype 6A (Shared) | 12553.06 [10072.11 to 15645.13] | 17476.24 [13999.28 to 21816.75]
  Serotype 6B (Shared): number analyzed (Participants) | 153 | 153
  Serotype 6B (Shared) | 9218.64 [7346.96 to 11567.14] | 14041.53 [11171.79 to 17648.42]
  Serotype 7F (Shared): number analyzed (Participants) | 155 | 155
  Serotype 7F (Shared) | 15451.96 [12500.49 to 19100.31] | 18039.04 [14593.41 to 22298.22]
  Serotype 9V (Shared): number analyzed (Participants) | 152 | 154
  Serotype 9V (Shared) | 3259.24 [2548.05 to 4168.93] | 5050.89 [3957.89 to 6445.73]
  Serotype 14 (Shared): number analyzed (Participants) | 154 | 155
  Serotype 14 (Shared) | 8486.72 [6720.27 to 10717.49] | 5719.04 [4521.91 to 7233.08]
  Serotype 18C (Shared): number analyzed (Participants) | 153 | 153
  Serotype 18C (Shared) | 7027.62 [5704.70 to 8657.32] | 5903.86 [4785.06 to 7284.24]
  Serotype 19A (Shared): number analyzed (Participants) | 155 | 156
  Serotype 19A (Shared) | 8441.43 [6620.55 to 10763.11] | 10834.58 [8499.57 to 13811.07]
  Serotype 19F (Shared): number analyzed (Participants) | 153 | 156
  Serotype 19F (Shared) | 4716.70 [3863.66 to 5758.07] | 3829.62 [3138.93 to 4672.28]
  Serotype 23F (Shared): number analyzed (Participants) | 153 | 153
  Serotype 23F (Shared) | 11319.82 [8635.69 to 14838.22] | 30686.58 [23314.40 to 40389.89]
  Serotype 22F (Unique to V114): number analyzed (Participants) | 156 | 144
  Serotype 22F (Unique to V114) | 5561.71 [3730.30 to 8292.26] | 35.68 [23.67 to 53.79]
  Serotype 33F (Unique to V114): number analyzed (Participants) | 154 | 152
  Serotype 33F (Unique to V114) | 19899.34 [14204.44 to 27877.46] | 1183.52 [844.22 to 1659.18]
Statistical Analysis 1: Comparison: V114 vs PCV13; Serotype 1: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.53, 95% CI 2-sided [0.38 to 0.75]
Statistical Analysis 2: Comparison: V114 vs PCV13; Serotype 3: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 1.62, 95% CI 2-sided [1.28 to 2.03]
Statistical Analysis 3: Comparison: V114 vs PCV13; Serotype 4: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.72, 95% CI 2-sided [0.57 to 0.93]
Statistical Analysis 4: Comparison: V114 vs PCV13; Serotype 5: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.86, 95% CI 2-sided [0.66 to 1.13]
Statistical Analysis 5: Comparison: V114 vs PCV13; Serotype 6A: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.72, 95% CI 2-sided [0.57 to 0.91]
Statistical Analysis 6: Comparison: V114 vs PCV13; Serotype 6B: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.66, 95% CI 2-sided [0.52 to 0.83]
Statistical Analysis 7: Comparison: V114 vs PCV13; Serotype 7F: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.86, 95% CI 2-sided [0.68 to 1.07]
Statistical Analysis 8: Comparison: V114 vs PCV13; Serotype 9V: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.65, 95% CI 2-sided [0.50 to 0.84]
Statistical Analysis 9: Comparison: V114 vs PCV13; Serotype 14: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 1.48, 95% CI 2-sided [1.16 to 1.90]
Statistical Analysis 10: Comparison: V114 vs PCV13; Serotype 18C: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 1.19, 95% CI 2-sided [0.95 to 1.48]
Statistical Analysis 11: Comparison: V114 vs PCV13; Serotype 19A: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.78, 95% CI 2-sided [0.60 to 1.01]
Statistical Analysis 12: Comparison: V114 vs PCV13; Serotype 19F: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 1.23, 95% CI 2-sided [1.00 to 1.52]
Statistical Analysis 13: Comparison: V114 vs PCV13; Serotype 23F: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 0.37, 95% CI 2-sided [0.28 to 0.49]
Statistical Analysis 14: Comparison: V114 vs PCV13; Serotype 22F: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 155.88, 95% CI 2-sided [101.84 to 238.59]
Statistical Analysis 15: Comparison: V114 vs PCV13; Serotype 33F: OPA GMT Ratio; Test type: Other — [test comment as in outcome 9, analysis 1]; GMT Ratio = 16.81, 95% CI 2-sided [11.74 to 24.08]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events: Up to 14 days after each vaccination, up to a total of 13.5 months; Serious adverse events: Approximately 1 month after Dose 4 (Up to 14 months); All-cause mortality: Up to 17 months
Description: The analysis population for deaths (all-causes) included all randomized participants. The analysis population for AEs included all randomized participants who received at least 1 dose of study vaccination.
Arm/Group | V114 | PCV13
All-Cause Mortality (participants affected / at risk) | 0/347 | 0/347
Serious Adverse Events (participants affected / at risk) | 24/347 | 23/346
Other Adverse Events (participants affected / at risk) | 340/347 | 340/346
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=347) | PCV13 (N=346)
Hamartoma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 3 (3) | 1 (2)
Milk allergy (Immune system disorders) | 1 (1) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 2 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Lymphadenitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Nephritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (5) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Kawasaki's disease (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=347) | PCV13 (N=346)
Diarrhoea (Gastrointestinal disorders) | 35 (43) | 20 (22)
Injection site erythema (General disorders) | 306 (878) | 309 (929)
Injection site induration (General disorders) | 281 (813) | 281 (787)
Injection site pain (General disorders) | 108 (178) | 83 (134)
Injection site swelling (General disorders) | 263 (670) | 276 (688)
Pyrexia (General disorders) | 227 (544) | 252 (610)
Nasopharyngitis (Infections and infestations) | 32 (34) | 37 (39)
Upper respiratory tract infection (Infections and infestations) | 20 (23) | 22 (29)
Decreased appetite (Metabolism and nutrition disorders) | 83 (132) | 84 (117)
Somnolence (Nervous system disorders) | 194 (430) | 190 (399)
Irritability (Psychiatric disorders) | 231 (522) | 210 (500)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 21 (23)
Eczema infantile (Skin and subcutaneous tissue disorders) | 18 (19) | 16 (16)
Erythema (Skin and subcutaneous tissue disorders) | 33 (44) | 31 (42)
Rash (Skin and subcutaneous tissue disorders) | 17 (21) | 18 (22)
Skin induration (Skin and subcutaneous tissue disorders) | 23 (29) | 18 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT04384107/Prot_001.pdf
  • Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT04384107/SAP_002.pdf